CLINICAL TRIAL: NCT03843658
Title: Identifying Novel Biomarkers in Early Rheumatology Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Arthritis Northwest PLLC (Industry)
Collaborators: Inova Diagnostics Inc (Unknown); Bristol-Myers Squibb (Industry); University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: R-18002
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Rheumatologic Disorder
MeSH Terms: conditions — Collagen Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Rheumatoid Arthritis: Clinician diagnosed rheumatoid arthritis
  Interventions: Other: There is no intervention, but a diagnosis.
- Spondyloarthropathy: Ankylosing spondylitis and psoriatic arthritis
  Interventions: Other: There is no intervention, but a diagnosis.
- Crystalline arthritis: Gout and Pseudo gout
  Interventions: Other: There is no intervention, but a diagnosis.
- Connective Tissue Disease: Lupus, myositis, scleroderma, and sjogren's
  Interventions: Other: There is no intervention, but a diagnosis.
- Non-Inflammatory arthritis: E.g. Osteoarthritis and Fibromyalgia
  Interventions: Other: There is no intervention, but a diagnosis.

INTERVENTIONS:
Other: There is no intervention, but a diagnosis. — Cohorts will be determined by the primary rheumatology diagnosis.

SUMMARY:
Patients new to a rheumatology practice will be asked if they want to consent to their blood sample, medical records, and hand/foot x-rays (with sharp scores) for the analysis and correlation with the diagnosis they will receive from the rheumatologist.

DETAILED DESCRIPTION:
At the end of their first visit new rheumatology patients will be asked for their interest in joining the Inova biomarker study. If yes, the patient will be consented, blood will be drawn for the Inova biomarkers, and x-rays will be sent for sharp scoring. Patients may decline and will not be part of the Inova study. Patients who decline will continue to receive standard of care treatment henceforth.

Patients in the Inova trial will receive a diagnosis from their doctor and are placed into separate cohorts based upon their diagnosis. The Inova biomarker results of each cohort will be cross-correlated with diagnoses, pre-screening tool results. Baseline disease activity and sharp scores will also be correlation variables.

ELIGIBILITY:
Inclusion Criteria:

* Newly referred Arthritis Northwest PLLC
* Age 18 or older

Exclusion Criteria:

* None.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All newly referred adults to Arthritis Northwest PLLC will be offered the opportunity to enroll in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-03-15 (Estimated); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
The correlation between novel biomarkers and the primary rheumatology diagnosis | 18 month enrollment period. No follow-up period
  Pearson's correlation coefficient of each biomarker to each cohort

IPD SHARING:
Plan to Share IPD: No